CLINICAL TRIAL: NCT04081194
Title: Cell Free Circulating Nucleic Acids as New Tumor Diagnostics From Human Plasma Samples.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Alameldin, Assisstent Lecturer, Assiut University
Other Study IDs: Sara Alameldin 20.06.2016
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: New Tumor Diagnostics From Human Plasma Samples

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group, Melanoma Patients: 15 patients of with Melanoma, Age between 40 and 90 years.
  -Withdrawal of Blood sample, Isolation of Exosomes:
  1. Bradford protein assay And Qubit protein assay.
  2. Bioanalyzer.
  3. Real time PCR.
- control group: 10 Persons without Melanoma, age > 40 years
  -Withdrawal of Blood sample, Isolation of Exosomes:
  1. Bradford protein assay And Qubit protein assay.
  2. Bioanalyzer.
  3. Real time PCR.

SUMMARY:
Cell Free Circulating Nucleic Acids as New Tumor Diagnostics From Human Plasma Samples.

DETAILED DESCRIPTION:
Cell free circulating free nucleic acids is new substrates for laboratory diagnostics in a number of medical areas including oncology, transfusion medicine, gynecology/obstetrics, inflammatory and autoimmune diseases etc.There are various qualities of cell free nucleic acids. In oncology, it has been shown that the early detection of cell free nucleic acids originating from the tumour preceeds the diagnostic detection of clinical relapse as done by imaging techniques or clinical symptoms by 6-8- months.

Exosomes are small, lipid bilayer membrane vesicles (30-100 nm) that are released from all cell types into the extracellular space. These tiny membrane vesicles transmit EV-mediated signals by proteins, lipids, nucleic acids and sugars, and the unique molecular pattern of this package direct the type of extracellular signal to be transmitted to target cells. Interest in exosomes range from their mode of action and various functions in the body to more practical applications such as development of biomarkers based on analysis of their RNA and protein content and their use in clinical diagnostics. It was proposed that micro RNAs are transferred through exosomes to recipient cells and can there mediate repression of their mRNA targets.

The use of highly expensive targeted therapies (e.g. tyrosine kinase inhibitors or PARP inhibitors) may become obsolete during therapy due to changes in the mutational molecular profile of the malignant tumour. Indeed, if early detection of cell free nucleic acids suggest therapy failure, new stratification of the patient and changed therapy modalities may be possible in the future, thus helping to prolong overall survival of tumour patients.

Aims of the Research:

* To isolate exosomes as a stable source of cell free nucleic acids.
* To perform protein profiling on the isolated exosomes.
* To isolate nucleic acids from exosomes for analysis.
* To define and develop standards and protocols for cell free nucleic acids analysis particularly regarding epigenetic alterations with emphasis on DNA methylation.
* Optimizing of pre-analytical process to improve the pre-analytical aspects of assays.
* To test the stability of methylated compared to non-methylated circulating DNA under various pre-analytical conditions.

ELIGIBILITY:
Inclusion Criteria:

* patients with Melanoma

Exclusion Criteria:

* patients with other types of malignancies

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study group: 15 Patients control Group: 10 Persons
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Isolation of Exosomes as a stable source of nucleic acid as an early Detection Method to diagnose Melanoma. | one year
  Real time PCR for detecting the presence of Melanoma relevant nucleic acids isolated of Exososmes.

CONTACTS AND LOCATIONS:
Overall Officials: Hesham A Abdel-Baset, Prof., Study Director — Assiut University- Faculty of Medicine- Clinical Pathology dept.
Locations (1):
- Assiut University Hospitals- Faculty of Medicine, Asyut, Egypt